CLINICAL TRIAL: NCT03619733
Title: Does Modified Heart Score Incorporating Undetectable and 99th Percentile High Sensitivity Troponin T Limits Improve Early, Safe Discharge for Suspected Acute Coronary Syndromes
Brief Title: Modified HEART as Rule Out for Suspected ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Royal Liverpool University Hospital (Other Government); University of Liverpool (Other)
Responsible Party: Principal Investigator, Aleem Khand, cosultant interventional cardiologist, Liverpool University Hospitals NHS Foundation Trust
Other Study IDs: AintreeNHS
Record Dates: First submitted 2018-07-01; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Chest Pain
Keywords: HEART score, troponins
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 123 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — this is an observational study. no intervention is planned

SUMMARY:
Validation of modified HEART score as a rule-out criterion for MACE at 6 weeks: a 2 centre prospective observational cohort with a direct comparison to TIMI, GRACE and high sensitive troponin T at limits of detection

Detailed description:

The HEART score, as defined previously by Backus et al1, is a risk score specifically developed for acute chest pain/ suspected acute coronary syndrome. The conventional scoring system for the troponin component of HEART is as follows: Troponin <99th percentile =0 (in the case of Hstn T [Roche} 14ng/l, 99th percentile up to X3 URL (99th percentile)= 1 (HSTN T =14-42ng/L, >x3 URN =2 (HSTN T >42ng/l).

We have previously defined that the optimal rule-out strategy for suspected acute coronary syndromes may well be a modified HEART score in a single centre study. This study is to prospectively validate the use of this score in a prospective unselected cohort of patients with possible acute coronary syndrome at 2 large secondary care centres

DETAILED DESCRIPTION:
Validation of modified HEART score as a rule-out criterion for MACE at 6 weeks: a 2 centre prospective observational cohort with a direct comparison to TIMI, GRACE and high sensitive troponin T at limits of detection

Detailed description:

The HEART score, as defined previously by Backus et al1, is a risk score specifically developed for acute chest pain/ suspected acute coronary syndrome. The conventional scoring system for the troponin component of HEART is as follows: Troponin <99th percentile =0 (in the case of Hstn T [Roche} 14ng/l, 99th percentile up to X3 URL (99th percentile)= 1 (HSTN T =14-42ng/L, >x3 URN =2 (HSTN T >42ng/l).

the investigators previously defined that the optimal rule-out strategy for suspected acute coronary syndromes may well be a modified HEART score in a single centre study. This study is to prospectively validate the use of this score in a prospective unselected cohort of patients with possible acute coronary syndrome at 2 large secondary care centres. The second centre (Royal Liverpool University Hospital) was external to where the initial cohort of 1642 patients were assessed that defined modified HEART as the optimal score.

The modified HEART score is as follows: HEART score can be re-calibrated (modified HEART) to undetectable hstnT and 99th percentile limits (<5= 0, ≥5-14=1, >14=2).

Troponin (HSTnT) Roche (elecsys) >14ng/l 2 5-14ng/l 1 <5ng/l 0

This 2 centre study will enrol consecutive patients with suspected acute coronary syndrome (defined as physician suspicion of ischaemic chest pain resulting in sampling of High sensitive troponin and undertaking an electrocardiogram at presentation).

For all troponin positive patients (HSTnT>14ng/l) the diagnosis will be adjudicated centrally with at least 2 'blinded' clinicians. The outcome will be MACE at 6 weeks. MACE will be defined by acute myocardial infarction, urgent or emergency coronary revascularisation and all cause death.

Power calculations (provided by clinical trials, university of Liverpool):

Assuming:

Prevalence of MACE events in the population with suspected ACS is 12.5% (as in MACROS) The anticipated sensitivity is 0.98 The acceptable value for the 95% confidence interval for sensitivity is 0.95 The power of the study is 80%

Then the number of events needed would be approximately 150. Thus 150/0.125 = 1200 suspected ACS admission would need to be enrolled

The study has been assessed by research boards at both hospitals and has been registered as an audit, with the primary aim of quality control of a novel accelerated chest pain pathway that has been recently implemented at both hospitals. The study does not require individualised patient consent and is supported by the Caldicott Guardian.

Secondary aims of the study are to compare the performance of modified HEART score with modified TIMI < or equal to 1 or 0 and modified GRACE score < or equal to 75 in terms of rule out for MACE at 6 weeks The investigators compare the 'performance' of modified HEART with the use of undetectable HSTnT <5ng/l (combined with a nonischaemic ECG). The latter is part of the recently adopted chest pain pathway at both recruiting hospitals with clear guidance of discharge at presentation for patients with chest pain who have an undetectable HSTnT and nonischaemic ECG. Therefore it will allow the research team to compare modified HEART virtual discharge with actual (rather than virtual) discharge for an approach based on undetectable HSTnT.

ELIGIBILITY:
Inclusion Criteria:consecutive presentations to A&E at 2 major urban hospital swith chest pain that the clinicans feel warrants a biomarker check for myocyte necrosis (high sensitive troponin) and presentation ECG

-

Exclusion Criteria:

primary presentation not chest pain

clear noncardiac cause of chest pain such as trauma life expectancy <1 year due to noncardiac pathology

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: consecutive presentations to A&E at 2 major urban hospital swith chest pain that the clinicans feel warrants a biomarker check for myocyte necrosis (high sensitive troponin) and presentation ECG
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of Major adverse cardiac event for patients with HEART score<=3 | 6 weeks
  adjudicated myocardial infarction, urgent or emergency coronary revascularisation, all-cause Death

SECONDARY OUTCOMES:
incidence of acute myocardial infarction for patients with HEART <=3 | 6 weeks
  adjudicated centrally by 2 physicans blinded to heart scores and to colleagues score

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Hospital Aintree, Liverpool
  - Royal Liverpool university hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khand AU, Backus B, Campbell M, Frost F, Mullen L, Fisher M, Theodoropoulos KC, Obeidat M, Batouskaya K, Carlton EW, Van Meerten K, Neoh K, Dakshi A, Mumma BE. HEART Score Recalibration Using Higher Sensitivity Troponin T. Ann Emerg Med. 2023 Oct;82(4):449-462. doi: 10.1016/j.annemergmed.2023.04.024. Epub 2023 Jun 10. PMID 37306637